CLINICAL TRIAL: NCT05506514
Title: Heat Therapy to Accelerate Muscle Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspetar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F202202032
Record Dates: First submitted 2022-04-24; First posted 2022-08-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Muscle Damage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hot (Experimental): 1h per day of water immersion at 42ºC for 11 days
  Interventions: Other: Water immersion
- Temperate (Sham Comparator): 30min per day of water immersion at 32ºC for 11 days
  Interventions: Other: Water immersion
- Cold (Experimental): 15min per day of water immersion at 15ºC for 11 days
  Interventions: Other: Water immersion

INTERVENTIONS:
Other: Water immersion — Comparison of 3 different water temperatures

SUMMARY:
The use of cold on muscle (Ice, Cold Water Immersion - CWI or cryotherapy) is a widespread practice used by health professionals, athletes or non-athletic population in the treatment of muscle soreness and soft tissue injuries. Application of cold on muscle is well known to decrease inflammation and reduce pain perception. However, some studies in humans and animals have reported contrasted effects of cold on muscle regeneration. On the other hand, recent studies in humans suggest that passive heat exposure can impact positively muscle protein synthesis, mitochondrial content and muscle torque in different types of populations. Rodent studies comparing heat and cold modalities following a muscle injury have reported that only repeated heat exposure enhances cross sectional area, accelerate macrophage infiltration in damaged fibers and enhances satellite cells activation which led to a faster muscle regeneration. As such heat therapy may be a promising tool to accelerate recovery after muscle injury. This study will investigate the effect of three distinct thermal interventions (Hot, Cold and Thermoneutral water immersion) on human skeletal muscle regeneration after an eccentric exercise. 36 participants will be distributed in a counterbalanced way into 3 groups being immersed for 15min to 1h per day in either HEAT or COLD or NEUTRAL water for 10 days following eccentric contractions.

DETAILED DESCRIPTION:
Background information & study rationale Cold exposure is a therapeutic modality supposed to enhance regeneration by alleviating pain, reducing tissue metabolism and restricting swelling and inflammation process. However, in light of some recent studies in animal models and in humans, cold application on injury might delay and impair muscle regeneration. At the same time, passive heat therapy emerges as a novel powerful strategy to enhance muscle recovery. Indeed, in healthy subjects it has been shown that 1H/day of passive heat exposure during 11 days enhances muscle torque through an improvement in contractile muscle function. In an immobilization context, it was recently reported that repeated passive heat exposure may reduce muscle atrophy and induce mitochondrial adaptations.

In rats, heat exposure following chemically-induced injury has been shown to enhance muscle regeneration by increasing muscle weight and cross-sectional area compared to non-heated or cold exposed rats. Macrophage infiltration were reported to migrate to injury site earlier in heated animals compared to non-heated and icing-treated groups. In the same way, heat exposure was associated with an increase in satellite cells number in injured muscle fibers. In addition, it has been shown that ice application immediately after injury has delayed the recovery of Myosin Heavy Chain (MyHC) profile and in contrast, repeated heat application has facilitated the recovery of an uninjured MyHC profile. Interestingly, collagen fibers area and TGF-β1 (a collagen precursors) were shown to be lower in heated groups than in control and iced groups suggesting less muscle fibrosis. Animal studies suggest that heat exposure may be a potent stimulus to enhance soft tissue regeneration after injury.

Very few human studies have examined the impact of local heat exposure on regeneration after muscle injury. A recent study focusing on muscle regeneration in humans, have investigated the effects of a heat therapy protocol composed of five daily 90 minutes sessions with heating garment performed after an exercise-based injury protocol composed of 300 maximal voluntary eccentric contractions. Compared to thermoneutral intervention, heated group presented a better recovery of strength in a fatigue resistance test consisting of 28 maximal isokinetic contractions at 180°/sec at 1 and 4 days after exercise session.

Study goals and objectives The goal of the present study is to determine the effect of multiple localized hot-water or cold-water immersions on muscle regeneration.

1. Principal research question/objective:

   - Determine if heat therapy can enhance and hasten muscle regeneration after an injury.
2. Secondary research questions/objectives (if applicable):

   * Clarify the usefulness of cold modalities to enhance muscle regeneration after an injury.
   * Investigate how heat and cold modalities influence biochemical markers of muscle regeneration.

Methodology & Project Duration The study will assess the effect of three distinct thermal therapies (Hot, Cold and Thermoneutral water immersion) on human skeletal muscle regeneration after a bout of electrically induced eccentric contractions. Participants will be assigned in a counterbalanced way to either HEAT or COLD or NEUTRAL group. Participants will be balanced after familiarization and baseline testing to ensure consistency between groups. Participants of all groups will complete a muscle injury protocol and will be treated with the assigned intervention immediately after injury and during the 10 following days.

Eccentric exercise protocol:

The eccentric exercise protocol will be inspired by the protocol conducted in several studies. This protocol (detailed below) is an exercise-based protocol that elicits substantially greater amounts of cytoskeletal damage compared with maximal voluntary contractions only. It allows us to better observe the impact of different therapies on the regeneration phases.

All participants will complete a familiarization week before the intervention. At the beginning of the intervention, baseline measurements will be tested for each participant involved in the study. The right leg will realize an electrically induced eccentric exercise protocol with the knee extensor muscles. The exercise protocol will consist of a total of 200 eccentric contractions: (i) 5 sets of 20 repetitions of eccentric leg extension at an angular velocity of 30°/second followed by (ii) 5 sets of 20 repetitions of eccentric leg extension at 180°/second using an isokinetic dynamometer (Biodex System 3). A 30 s break between each set and a 5 min break between the slow and fast contractions will be given. All muscle contractions will be induced by electrical stimulations (ES) without any voluntary contribution. Impulse trains (200 μs single pulse duration; 40 Hz; maximal current, 100 mA) will be delivered under manual control over two stimulation electrodes placed across the vastus lateralis muscle of the assigned leg; 5 cm from the top of the patella and; 5 cm from the anterior superior iliac spine. The subjects will be carefully instructed not to produce any voluntary muscle contraction during this phase of the exercise protocol. Electrical stimulation will begin at the initiation of downward movement of the dynamometer lever arm, and it will be turned off at the end of this downward movement. Range of motion during the eccentric exercise measurement will be set from 90° to 10°.

Thermal interventions:

Local heating, local cooling and sham intervention will be applied by immersing the legs up to the waist in a water bath. Thermal interventions will be applied 11 times during the protocol. They will be initiated 1 hour (D0) after the completion of eccentric exercise protocol and every day for 10 days (D1-2-3-4-5-6-7-8-9-10). Heat intervention (HOT) will consist of immersing the legs for 60 minutes in a hot water bath maintained at a temperature of 42°C. Cold intervention (COLD) will consist of immersing the legs for 15 minutes in a cold-water bath maintained at a temperature of 15°C. For the sham intervention (NEUTRAL), participant legs will be immersed for 30 minutes in a thermoneutral water bath maintained at a temperature of 32°C. Thermal interventions from day 1 to day 10 will be performed each day immediately after the completion of daily testing measurement.

Quadriceps muscle temperature will be monitored (during day 3) using a needle thermo-sensor. This measure aims to identify the changes in muscle temperature induced by each bath temperature at different muscle depth. The needle will be inserted to a depth of 2.5cm into the vastus lateralis of the treated leg after local anesthesia of the skin (2 mL of Xylocaine without adrenaline). Core temperature will be monitored using ingestible pills thermometer (e-Celcius, Bodycap, France). Room temperature will be set at 24° and 40% humidity to not interfere with treatment effects.

Familiarization visit:

A familiarization visit will be completed during the month preceding the baseline measurements. It will be composed of an eccentric exercise initiation protocol with 4 electrically induced eccentric contractions of quadriceps muscle at 30°/second and 4 at 180°/second. Participants will also experience a lightened version of the neuromuscular tests (4 peak twitch contractions, 3 maximal voluntary contractions, 2 EMG measurements, 5 RFD contractions, 5 contractions at 120°/second) in order to accustomed them to the testing procedure. During the familiarization visit, a consent form and a Par-Q questionnaire will also be completed and an anthropometric analysis (ISAK) will be realised by participants.

Data collection procedure:

All the tests from day 1 to day 10 will be realized before the thermal intervention to avoid any acute effect.

Complete neuromuscular testing:

A complete neuromuscular test battery will be performed at baseline (i.e. the week preceding the beginning of the intervention) and post-injury at day 10. It will be composed of an electrically evoked twitch measure, 3 maximal voluntary contractions in isometric mode, 5 contractions to assess rate of force development, an electromyographic analysis, a shear wave elastography analysis, a fatigue test and a muscle soreness evaluation of the vastus lateralis.

Intermediate neuromuscular testing:

An Intermediate neuromuscular testing will be performed at day 2 and day 4 after the eccentric exercise. The intermediate test battery will only include the electrically evoked twitch measure, 3 maximal voluntary contractions in isometric mode, 5 contractions to assess RFD, an electromyographic analysis, a shear wave elastography analysis and a muscle soreness evaluation of the vastus lateralis.

Simplified neuromuscular testing:

A simplified neuromuscular testing will be performed at day 1, 2, 3 and then every day from day 5 to day 9. It will only be composed of an electrically evoked twitch measure and a muscle soreness evaluation of the vastus lateralis.

Muscle biopsy sampling:

Biopsies of the vastus lateralis will be taken at baseline (i.e. the week preceding the beginning of the intervention) and on day 5 and 11. The biopsy taken the baseline measurement will be sampled on the contralateral leg.

Thermal imaging:

Thermal imaging of the legs will be recorded each day from day 1 to day 10 before the completion of any neuromuscular tests or biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Adult (18 to 45 yrs)
* Physically active

Exclusion Criteria:

* Contraindication to physical activity as per the Par-Q questionnaire
* Neural, skin or muscular pathology.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength after 2 days | 2 days post exercise
  Change in maximal knee extensor isometric voluntary force (kg) 2 days after the exercise as compared to baseline
Change in muscle strength after 4 days | 4 days post exercise
  Change in maximal knee extensor isometric voluntary force (kg) 4 days after the exercise as compared to baseline
Change in muscle strength after 10 days | 10 days post exercise
  Change in maximal knee extensor isometric voluntary force (kg) 10 days after the exercise as compared to baseline

SECONDARY OUTCOMES:
Change in muscle fiber | 5 days post exercise
  Change in the proportion of centrally nucleated muscle fiber (%) in a muscle biopsy of the vastus lateralis at 5 days post exercise as compared to baseline
Change in muscle fiber | 11 days post exercise
  Change in the proportion of centrally nucleated muscle fiber (%) in a muscle biopsy of the vastus lateralis at 11 days post exercise as compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Aspetar sport medicine hospital, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: No
No personal identifier will be shared. All data will be anonymous

REFERENCES:
- [Background] Dablainville V, Mornas A, Normand-Gravier T, Al-Mulla M, Papakostas E, Olory B, Fermin TM, Zampeli F, Nader N, Alhammoud M, Bayne F, Sanchez AMJ, Cardinale M, Candau R, Bernardi H, Racinais S. Muscle regeneration is improved by hot water immersion but unchanged by cold following a simulated musculoskeletal injury in humans. J Physiol. 2025 Dec;603(23):7603-7625. doi: 10.1113/JP287777. Epub 2025 May 28. PMID 40437768